CLINICAL TRIAL: NCT05179473
Title: Changing Practice: Prognosis and Diagnosis of Spasticity in Acute-post Stroke Patients: a Pilot Study
Brief Title: Prognosis and Diagnosis of Spasticity in Acute-post Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Mindy F. Levin, Professor, McGill University
Other Study IDs: MP-37-2019-5298
Record Dates: First submitted 2021-12-10; First posted 2022-01-05 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Stroke, Acute; Stroke, Ischemic; Stroke Hemorrhagic; Spasticity as Sequela of Stroke
Keywords: stroke; spasticity; imaging; prognosis; diagnosis; upper limb; lower limb
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Muscle Spasticity; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute stroke patients: 12 weekly evaluations starting within the first week post-stroke. Follow-up assessment at week 16. MRI at week 6.

SUMMARY:
Spasticity, or greater muscle resistance, is a major disabling condition following stroke. Recovery of lost motor function in patients with stroke may be affected by spasticity, which most commonly develops in elbow and ankle muscles. However, despite its clinical relevance, the natural development of spasticity over the first 3 months after stroke is not clearly understood. Indeed, common clinical measures of spasticity such as the Modified Ashworth Scale (MAS) do not take into account the neurophysiological origin of spasticity and lack reliability and objectivity.

The objective of this study is to examine the natural history of the development of spasticity among patients with stroke over the first 3 months using a new neurophysiological measure (TSRT, the tonic stretch reflex threshold angle) and its velocity sensitivity (mu) in comparison to MAS and other common clinical tests. In addition, detailed brain imaging will be used to understand the relationship between damage to brain regions relevant to the development of spasticity and TSRT/mu values.

It is hypothesized that 1) TSRT/mu will indicate the presence of spasticity earlier than MAS/clinical tests; 2) TSRT/mu measures will be more closely related to motor impairments and activity limitations than MAS; 3) the lesion severity (identified by imaging) will be related to the change in TSRT/mu values.

Outcomes will be measured in a pilot cohort of 12 patients hospitalized for first-ever stroke. Measurements will be taken at the bedside within the 1st week of the patient's admission and will be done once per week for 12 weeks with a follow-up at week 16. Brain Imaging will be done around the 6th week post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke in Middle Cerebral Artery area resulting in hemiparesis.
* Hemorrhagic or ischemic
* Medically stable
* Able to provide informed consent

Exclusion Criteria:

* Severe cognitive disorders
* Ataxia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from acute care facilities such as general hospitals and stroke units in Montreal area hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
TSRT | up to 16 weeks
  Tonic stretch reflex threshold measured in the elbow flexors or ankle plantarflexors
Mu | up to 16 weeks
  Velocity sensitivity of the TSRT
Modified Ashworth Scale (MAS) | up to 16 weeks
  Measure of the increase of muscle resistance to stretch felt by examiner in the elbow flexors or ankle plantarflexors
Reflexes | up to 16 weeks
  Measured in the elbow flexors or ankle plantarflexors

SECONDARY OUTCOMES:
Active Range of Motion (AROM) | up to 16 weeks
  Measured in elbow or ankle for flexion and extension
Passive Range of Motion (PROM) | up to 16 weeks
  Measured in elbow or ankle for flexion and extension
Semmes-Weinstein filaments | up to 16 weeks
  Measure of the sensory threshold in index and thumb or first toe and middle-plantar surface of the foot
Maximal Voluntary Force (MVF) | up to 16 weeks
  Measured in the elbow flexors and extensors, and in the ankle dorsiflexors and plantarflexors
Fugl-Meyer Assessment Upper Limb/Lower Limb (FMA - UL/LL) | up to 16 weeks
  Assessment of motor function, balance, sensation and joint function in the upper and lower limb
Berg Balance Scale | up to 16 weeks
  Measure of balance in standing
Box and Blocks Test (BBT) | up to 16 weeks
  Number of blocks moved by the more-affected arm compared to the less-affected arm
Timed Up and Go (TUG) | up to 16 weeks
  Activity measure of whole body function

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Wein, MD, Principal Investigator — Montreal Neurological Institute; Alexander Thiel, MD, Study Chair — Jewish General Hospital - McGill University; Marie-Helene Boudrias, PT, PhD, Study Chair — McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No